CLINICAL TRIAL: NCT01171144
Title: Time Trend Analysis of Diarrhoea-related Incidence, Hospitalizations, and Deaths in Children < 5 Years of Age in Panama by Monitoring Secondary Data Sources From 1990-2010
Brief Title: Trends Over Time (1990-2010) of Diarrhoea-related Incidence, Hospitalizations and Deaths in Children of Panama
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111757
Record Dates: First submitted 2010-07-15; First posted 2010-07-28 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: None Retained — No samples are retained.

GROUPS / COHORTS (1):
- Gastroenteritis Group: All children suffering with gastroenteritis
  Interventions: Other: Epidemiologic Surveillance System of the Ministry of Health of Panama; Other: Mortality database of the Contraloria General de la Republica; Other: Hospital discharge records

INTERVENTIONS:
Other: Epidemiologic Surveillance System of the Ministry of Health of Panama — Reviewing the Epidemiologic Surveillance System of the Ministry of Health of Panama
Other: Mortality database of the Contraloria General de la Republica — Reviewing the Mortality database of the Contraloria General de la Republica
Other: Hospital discharge records — Reviewing the hospital discharge records

SUMMARY:
This study aims at collecting data from secondary sources to obtain baseline incidence and monitor trends over time (1990 - 2010) of reported gastroenteritis cases, gastroenteritis related hospital discharges and gastroenteritis related deaths in children < 5 years of age in Panama before and after implementation of Rotarix™ universal mass vaccination.

DETAILED DESCRIPTION:
Data will be collected from systematic review of the databases of epidemiologic surveillance system, hospital discharges and deaths for all cause gastroenteritis related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diarrhea cases, diarrhea associated hospital discharges, and diarrhea related deaths occurring in children <5 years of age during the period analyzed and registered in the Epidemiologic Surveillance System of the Ministry of Health, in the mortality database of the Contraloría General de la República and in the hospital discharge records of the selected hospitals, will be collected for the study.

Exclusion Criteria:

* Not applicable

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children <5 years of age reported with gastroenteritis, gastroenteritis related hospital discharges and gastroenteritis related deaths in Panama, between 1990 and 2010.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of all cause reported gastroenteritis | In post vaccine introduction period (2006-2010) compared to pre-vaccination period (1990-2005)
Occurrence of all cause gastroenteritis related hospital discharges | In post vaccine introduction period (2006-2010) compared to pre-vaccination period (2000-2005)
Occurrence of all cause gastroenteritis related deaths. | In post vaccine introduction period (2006-2010) compared to pre-vaccination period (1990-2005)

SECONDARY OUTCOMES:
Occurrence of all cause gastroenteritis-related cases by year, age groups and region | From 1990 to 2010
Occurrence of all cause gastroenteritis related hospital discharge by year, age groups, hospital and setting | From 2000 to 2010
Occurrence of all cause gastroenteritis related deaths by year, age groups and region | From 1990 to 2010

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Panama City, Panama